CLINICAL TRIAL: NCT00840281
Title: A Relative Bioavailability Study of Cefprozil 500 mg Tablets Under Fasting Conditions
Brief Title: Cefprozil 500 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B036556
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-07-21 (Estimated); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Cefprozil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Cefprozil 500 mg Tablets
- 2 (Active Comparator)
  Interventions: Drug: Cefzil® 500 mg tablets

INTERVENTIONS:
Drug: Cefzil® 500 mg tablets — 1 x 500 mg, single-dose fasting
  Arms: 2
Drug: Cefprozil 500 mg Tablets — 1 x 500 mg, single-dose fasting
  Arms: 1

SUMMARY:
The objective of this study is to compare the relative bioavailability of cefprozil 500 mg tablets (Teva Pharmaceuticals USA) with that of Cefzil® 500 mg tablets (Bristol-Myers Squibb) in healthy, non-smoking adults under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Subjects selected for this study will be non-smokers at least 18 years of age. Subjects will have a BMI (body mass index) of 30 or less.
* Each subject shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history.
* Each female subject will be given a serum pregnancy test as part of the pre-study screening process.
* At the end of the study, the subjects will have an exit evaluation consisting of interim history, global evaluation, and clinical laboratory measurements.
* Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the trial for clinical laboratory measurements.
* Clinical laboratory measurements will include the following.

  * HEMATOLOGY: hematocrit, hemoglobin, WBC count with differential, RBC count, platelet count
  * CLINICAL CHEMISTRY: creatinine, BUN, glucose, SGOT/AST, SGPT/ALT, bilirubin, and alkaline phosphatase
  * HIV antibody, hepatitis B surface antigen, hepatitis C antibody screens
  * URINE ANALYSIS: pH, specific gravity, protein, glucose, ketones, bilirubin, occult blood, and cells
  * Drugs of Abuse Screen

Exclusion Criteria:

* Subjects with a significant recent history of chronic alcohol consumption (past 2 years), drug addiction, or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma (past 5 years), diabetes, psychosis or glaucoma will not be eligible for this study.
* Subjects whose clinical laboratory test values are greater than 20% outside the normal range may be retested. If the clinical values are outside the range on retesting, subjects will not be eligible to participate in the study unless the clinical investigator deems the results to not be significant.
* Subjects who have a history of allergic responses to the class of drug being tested will be excluded from the study.
* Subjects who use tobacco in any form will not be eligible to participate in the study. Three months abstinence is required.
* All subjects will have urine samples assayed for the presence of drugs of abuse as part of the clinical laboratory screening procedures and at each dosing period check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate.
* Subjects should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study.
* Subjects who have taken any investigational drug within thirty (30) days prior to the first dosing of the study will not be allowed to participate.
* Female subjects who are pregnant, breast-feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain froom sexual intercourse or use a reliable barrier method (e.g. condom, IUD) of contraception during the course of the study (first dosing until last blood collection) or they will not be allowed to participate. Female subjects who have used hormonal oral contraceptives within 14 days of dosing or implanted or injected hormonal contraceptives within 180 days of dosing will not be allowed to participate.
* All female subjects will be screened for pregnancy at check-in each study period. Subjects with positive or inconclusive results will be withdrawn from the study.
* Subjects who do not tolerate venipuncture will not be allowed to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2003-09; Primary Completion 2003-09 (Actual); Study Completion 2003-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Parham, M.D., Principal Investigator — Gateway Medical Research
Locations (1):
- Gateway Medical Research, Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cefprozil (Test) First: 500 mg Cefprozil Tablets test product dosed in first period followed by 500 mg Cefzil® Tablets reference product dosed in the second period.
- Cefzil® (Reference) First: 500 mg Cefzil® Tablets reference product dosed in first period followed by 500 mg Cefprozil Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Cefprozil (Test) First | Cefzil® (Reference) First
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Cefprozil (Test) First | Cefzil® (Reference) First
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Cefprozil (Test) First | Cefzil® (Reference) First
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cefprozil (Test) First | Cefzil® (Reference) First | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 19 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 13 | 11 | 24
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 0 | 1 | 1
  Black | 4 | 1 | 5
  White | 15 | 17 | 32
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 38

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 12 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Cefprozil (Test): 500 mg Cefprozil Tablets test product dosed in either period.
- Cefzil® (Reference): 500 mg Cefzil® Tablets reference product dosed in either period.
Arm/Group | Cefprozil (Test) | Cefzil® (Reference)
Number analyzed (Participants) | 38 | 38
ng/mL | 11.509 (3.314) | 11.573 (3.48)
Statistical Analysis 1: Comparison: Cefprozil (Test) vs Cefzil® (Reference); Test type: Non-Inferiority or Equivalence — The ANOVA model containing factors for sequence of products, subjects within sequence, periods, and products was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 100, 90% CI [94.9 to 105] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 12 hour period.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefprozil (Test) | Cefzil® (Reference)
Number analyzed (Participants) | 38 | 38
ng*h/mL | 34.528 (10.625) | 34.033 (9.471)
Statistical Analysis 1: Comparison: Cefprozil (Test) vs Cefzil® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101, 90% CI [98.6 to 103] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 12 hour period.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cefprozil (Test) | Cefzil® (Reference)
Number analyzed (Participants) | 38 | 38
ng*h/mL | 34.890 (10.727) | 34.379 (9.515)
Statistical Analysis 1: Comparison: Cefprozil (Test) vs Cefzil® (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101, 90% CI [98.7 to 103] — [estimate comment as in outcome 1, analysis 1]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.